CLINICAL TRIAL: NCT04346459
Title: Evaluation of Three Different Techniques for Tracheal Intubation Via Supraglottic Airway Devices: A Comparative Randomised Study
Brief Title: Three Different Techniques for Tracheal Intubation Via Supraglottic Airway Devices
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital of Patras (Other)
Responsible Party: Principal Investigator, Maria Spyraki, Principal Investigator, University Hospital of Patras
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 11/11/2019anesthesia
Record Dates: First submitted 2020-04-10; First posted 2020-04-15 (Actual); Last update posted 2023-07-03 (Actual); Status verified 2023-06

CONDITIONS: Tracheal Intubation
Keywords: tracheal intubation; supraglottic airway device

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group A- Fastrach (control group) (Active Comparator): Group of 40 patients scheduled for elective surgery under general anesthesia are planned to be intubated using intubating laryngeal mask airway "Fastrach" following blind intubating method through "Fastrach"
  Interventions: Procedure: Tracheal intubation through "Fastrach" - Group A
- Group B- I-gel (Active Comparator): Group of 40 patients scheduled for elective surgery under general anesthesia are planned to be intubated using "I-gel" supraglottic airway device as a conduit for tracheal intubation guided by a fiberoptic bronchoscope.
  Interventions: Procedure: Tracheal intubation through "I-gel" - Group B
- Group C- Protector (Active Comparator): Group of 40 patients scheduled for elective surgery under general anesthesia are planned to be intubated using the "Protector" laryngeal mask airway as a conduit for tracheal intubation guided by a fiberoptic bronchoscope.
  Interventions: Procedure: Tracheal intubation through "Protector" - Group C

INTERVENTIONS:
Procedure: Tracheal intubation through "Fastrach" - Group A — Insertion of the intubating laryngeal mask "Fastrach" and blind tracheal intubation through the device
  Arms: Group A- Fastrach (control group)
Procedure: Tracheal intubation through "I-gel" - Group B — Insertion of the supraglottic airway device "i-gel" and tracheal intubation through the device guided by a fiberoptic bronchoscope
  Arms: Group B- I-gel
Procedure: Tracheal intubation through "Protector" - Group C — Insertion of the laryngeal mask "Protector" and tracheal intubation through the device guided by a fiberoptic bronchoscope
  Arms: Group C- Protector

SUMMARY:
This study compares three different supraglottic airway devices used as a conduit for tracheal intubation in order το determine which one achieves the highest success rate of first attempt intubation

DETAILED DESCRIPTION:
Prospective, randomized, comparative, clinical, controlled study, that is approved by the Ethics Commitee of the University of Patras (10.12.2019) and takes part in the University Hospital of Patras. Depending on the supraglottic airway device (SGA)/ laryngeal mask airway (LMA) used to achieve intubation (Fastrach, I-gel, Protector), partcipants will be randomly allocated into three groups; Group A, B and C (Fastrach, I-gel, Protector respectively).

In the preoperative setting, a complete preanesthetic evaluation will be performed, including a detailed airway assessment (prediction of difficulty in face mask ventilation, insertion of SGA/LMA and intubation).

All patients are scheduled to undergo an elective surgery under general anesthesia. Before induction, all patients will be preoxygenated with FiO2 100% for at least 5 minutes. After induction, using rocuronium 0.6mg/kg to facilitate neuromuscular blockade, face mask ventilation follows.

1. Group A- Fastrach: The intubating laryngeal mask airway (Fastrach) will be placed to the patients of this group. After the mask is correctly placed and patients are adequately ventilated, they will be intubated through the mask using its own endotracheal tube according to the blind technique insertion.
2. Group B- I-gel: The supraglottic airway device (I-gel) will be placed to the patients of this group. After the mask is correctly placed and patients are adequately ventilated, they will be intubated through the mask using a fiberoptic bronchoscope to guide endotracheal tube's placement.
3. Group C- Protector: The supraglottic airway device (Protector) will be placed to the patients of this group. After the mask is correctly placed and patients are adequately ventilated, they will be intubated through the mask using a fiberoptic bronchoscope to guide endotracheal tube's placement.

In all groups (A, B, C) up to 3 attempts of SGA/LMA placement and up to 3 attempts of intubation are allowed to be made.

In case of an emerging unpredicted difficult airway and a concurrent unsuccessful SGA/LMA placement, then the algorithm of the difficult airway will be immediately followed. Video-assisted laryngoscopy will be the first option rescue alternative.

The time of the whole procedure from the beginning of SGA's/LMA's placement effort until the successful intubation will be recorded, along with the evaluation of the success rate of first intubation attempt.

ELIGIBILITY:
Inclusion Criteria:

* Patients (age ≥ 18 yrs) scheduled for an elective surgery under general anesthesia
* Written informed consent to participate in the trial

Exclusion Criteria:

* Age < 18 yrs
* Non- elective (urgent/ emergency) procedures or multi-trauma patients
* Obstetric population
* Surgery performed under regional anesthesia
* Contraindication to LMA insertion
* Predicted difficulty in LMA insertion (at least one out of four "RODS" criteria)
* Contraindication to the use of neuromuscular blockade or situations that require spontaneous breathing
* Indication for awake intubation or surgical airway
* Patients' involvement in another clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2020-01-10 (Actual); Primary Completion 2023-03-23 (Actual); Study Completion 2023-03-23 (Actual)

PRIMARY OUTCOMES:
Success rate of intubation at first attempt | Up to study completion, an average of 2 years
  Recording of successful tracheal intubation at first attempt (yes/no) and evaluation of the success rate at first attempt

SECONDARY OUTCOMES:
Time required for tracheal intubation | Up to study completion, an average of 2 years
  Time required from the beginning of the insertion of the supraglottic airway device/ laryngeal mask until the endotracheal tube is successfully placed confirmed by continuous waveform capnography (3 cycles)
Time required for successful supraglottic airway device/ laryngeal mask placement | Up to study completion, an average of 2 years
  Time required from the beginning of the insertion of the supraglottic airway device/ laryngeal mask until adequate ventilation is confirmed by continuous waveform capnography (3 cycles)

CONTACTS AND LOCATIONS:
Overall Officials: Gregorios Voyagis, MD, PhD, Study Chair — University of Patras, Department of Anesthesiology and Critical Care
Locations (1):
- University Hospital of Patras, Pátrai, Achaia, Greece